CLINICAL TRIAL: NCT04306978
Title: Impact of the CareLink Express Remote Monitoring System on Early Detection of Atrial Fibrillation and Cardiovascular Risk Reduction in Patients With Implantable Cardiac Pacemakers
Brief Title: Impact of the CareLink Express Remote Monitoring System on Early Detection of Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Research Institute for Complex Problems of Cardiovascular Diseases, Russia (Other)
Responsible Party: Principal Investigator, Sergey Mamchur, Head of Department of Diagnosis of Cardiovascular Diseases, Research Institute for Complex Problems of Cardiovascular Diseases, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0546-2015-0017
Record Dates: First submitted 2018-12-23; First posted 2020-03-13 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; tromboembolism; remote monitoring
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CareLink Express RM system (Active Comparator): Patients in the remote monitoring (RM) group will undergo the implantation of Ensura DR MRI SureScan pacing system. Patients in the RM group should visit the main follow-up clinic 12 weeks after discharge, and then the device data will be remotely transmitted to the CareLink Express Network at least once in 3 months. Research personnel will contact patients by telephone once in 6 months. If participants indicate they have experienced a study outcome event (corresponding to the study endpoints), the event will be recorded. If remote transmission or telephone call data require to make clinical decision an in-hospital visit will be induced.
  Interventions: Other: CareLink Express RM system
- Standard follow-up (Active Comparator): Patients in the control group will receive Adapta DR pacing system without remote monitoring using. All patients from the control group should have the first in-hospital visit 12 weeks after pacemaker implantation. Then, the follow-up will be provided according to the standard guidelines
  Interventions: Other: Standard follow-up

INTERVENTIONS:
Other: CareLink Express RM system — CareLink Express remote monitoring system consists of implantable pacemaker CareLink Express station for implanted Medtronic cardiac devices and provides remote data transmissions
  Arms: CareLink Express RM system
Other: Standard follow-up — Follow-up will be provided according to the standard guidelines (HRS/EHRA Expert Consensus on the Monitoring of Cardiovascular Implantable Electronic Devices (CIEDs): Description of Techniques, Indications, Personnel, Frequency and Ethical Considerations; 2008)
  Arms: Standard follow-up

SUMMARY:
The study results will be used to check the hypothesis that CareLink Express remote monitoring system increases the detection rate of asymptomatic AF and allows to change timely the treatment strategy in patients at high risk of thromboembolic events, e.g. anticoagulation therapy onset, electrical cardioversion or/and PVI.

DETAILED DESCRIPTION:
It is expected to enroll 200 consecutive patients without previously diagnosed AF, who have indications for implantation of dual chamber cardiac pacemakers according to the current guidelines. All the patients will be randomly assigned into 2 groups. Patients in the RM group will undergo the implantation of Ensura DR MRI SureScan pacing system, whereas patients in the control group will receive ADAPTA DR pacing system without RM using. The impact of the Care Link Express service on prevention of thromboembolism will be evaluated. The rate of in-hospital visits for 1 patient per year and compliance with scheduled CareLink transmissions (ratio of the number of the performed transmissions to the planned ones) will be assessed in all patients in the remote monitoring group. Moreover, we are going to estimate the interaction between the follow-up center and other healthcare facilities equipped with the CareLink Express service, which will facilitate faster treatment decision.

ELIGIBILITY:
Inclusion Criteria:

* patients with indications for implantation of dual chamber cardiac pacemaker
* patients with no AF history;
* written informed consent.

Exclusion Criteria:

* patients with contraindications for CIED implantation;
* patients with previously implanted CIEDs;
* infection;
* patients with previously diagnosed AF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-09-21 (Actual); Primary Completion 2022-09-21 (Estimated); Study Completion 2023-01-21 (Estimated)

PRIMARY OUTCOMES:
time (days) from the pacemaker system implantation to the first AF episode detected by ESG or EGM | 24 months
  the episode should be evaluated by the follow-up clinic physician(s) and meet the appropriate criteria (irregular RR intervals and distinct P waves, ≥30s episode duration)

SECONDARY OUTCOMES:
thromboembolic events | 24 months
  Number of participants with ischaemic stroke, transient ischaemic attack and thromboembolism (including any arterial embolism and paradoxical embolism)
hospitalization for cardiovascular events | 24 months
  Number of participants with arrhythmia, heart failure decompensation, thromboembolic events
the number of non-planned induced visits in the follow-up center | 24 months
  Number of visits for 1 patient per year
correction in the medical therapy | 24 months
  Number of participants with antiarrhythmic therapy or/and oral anticoagulation therapy initiated after the AF detection
cardioversion | 24 months
  Number of patinents underwent electrical cardioversion
catheter/surgical PVI | 24 months
  Number of patients underwent catheter or surgical atrial fibrillation ablation
all-cause mortality | 24 months
  Number of patients dead because of all causes

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute for Complex Problems of Cardiovascular Diseases, Kemerovo, Russia

IPD SHARING:
Plan to Share IPD: Undecided